CLINICAL TRIAL: NCT05085275
Title: Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Determine the Effect of Ferric Citrate on Time to a Composite Endpoint of Initiation of Maintenance Dialysis or All-cause Mortality vs Placebo in Adults With Advanced CKD
Brief Title: Ferric Citrate for the Prevention of Renal Failure in Adults With Advanced Chronic Kidney Disease
Acronym: FRONTIER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: USRC Kidney Research (Network)
Collaborators: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USRC-2021-002
Record Dates: First submitted 2021-10-06; First posted 2021-10-20 (Actual); Results first posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-04

CONDITIONS: Anemia, Iron Deficiency; Hyperphosphatemia; Renal Insufficiency, Chronic; Renal Anemia; Disease Progression; Cardiovascular; Iron
Keywords: ferric citrate
MeSH Terms: conditions — Anemia, Iron-Deficiency; Hyperphosphatemia; Renal Insufficiency, Chronic; Disease Progression | interventions — ferric citrate

STUDY DESIGN:
Intervention Model Description: Randomized, placebo controlled, double-blind, parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ferric citrate (Experimental): Supplied as tablets for oral administration containing 1 gram ferric citrate (210 milligrams of ferric iron). Administered orally with meals or snacks.
  Interventions: Drug: Ferric Citrate 1 GM Oral Tablet [AURYXIA]
- Placebo (Placebo Comparator): Tablets, matching in color and size to ferric citrate.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ferric Citrate 1 GM Oral Tablet [AURYXIA] — All subjects will be instructed to take study drug (ferric citrate or placebo) at a fixed dose of 2 tablets per meal or snacks, up to three times per day. The maximum dose is 6 tablets per day. No additional tablets (beyond a total of 6 per day) should be taken. Tablets should not be crushed or chewed.
  Other Names: Auryxia
  Arms: Ferric citrate
Drug: Placebo — All subjects will be instructed to take study drug (ferric citrate or placebo) at a fixed dose of 2 tablets per meal or snacks, up to three times per day. The maximum dose is 6 tablets per day. No additional tablets (beyond a total of 6 per day) should be taken. Tablets should not be crushed or chewed.
  Arms: Placebo

SUMMARY:
A 9-month randomized, double-blind, placebo-controlled study to compare the effect of fixed dose ferric citrate versus placebo in patients with advanced chronic kidney disease (eGFR ≤20 ml/min/1.73m2) on the composite endpoint of time to initiation of maintenance dialysis or all-cause mortality.

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind, placebo-controlled clinical trial is being conducted to determine the effect of ferric citrate on the time to a composite endpoint of initiation of maintenance dialysis or all-cause mortality in patients with non-dialysis dependent, advanced CKD. Up to 400 subjects will be randomized in 1:1 ratio to receive either ferric citrate or matching placebo. All subjects will initiate dosing at 2 tablets per meal or snacks, up to 3 times per day (maximum of 6 tablets per day). The dose of ferric citrate/placebo will only be adjusted based on safety and/or tolerability. Given the double-blind design of this trial, investigators will be instructed to not prescribe commercial Auryxia to either study arm. Study visits during the treatment period are to be conducted as part of routine scheduled clinical encounters. Standard of care local laboratory results will be collected however no study specific laboratory tests other than a pregnancy test in women of child-bearing potential will be required.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients greater or equal to 18 years old.
2. Diagnosis of NDD advanced CKD, regardless of etiology. Advanced CKD is defined as at least one local laboratory determined estimated glomerular filtration rate (eGFR) ≤20 ml/min/1.73m2 (calculated per any commonly used method or equation for estimating eGFR) within 90 days of Day 1.
3. Most recent transferrin saturation (TSAT) less than or equal to 45% within 45 days of Day 1.
4. Most recent serum phosphate is greater or equal to 3.0 mg per dL within 45 days of Day 1.
5. Most recent ferritin is less than or equal to 500 ng per mL within 45 days of Day 1.
6. Women of child-bearing potential must have a negative serum or urine pregnancy test within 28 days prior to Day 1.
7. Understands the procedures and requirements of the study and provides written informed consent and authorization for protected health information disclosure.

Exclusion Criteria:

1. Patients who, in the opinion of the Investigator, have acute kidney injury rather than CKD.
2. Patients with planned/imminent maintenance dialysis, or that are anticipated to begin maintenance dialysis within 8 weeks from Screening, in the opinion of the Investigator.
3. A known allergy or intolerance to ferric citrate or any of its constituents.
4. Hypersensitivity reaction to previous oral iron therapy.
5. History of hemochromatosis or iron overload syndrome (e.g., hereditary sideroblastic anemia, thalassemia, polycythemia vera).
6. Active malignancy requiring current treatment except for non-melanoma skin cancer regardless of treatment.
7. Active drug or alcohol dependence or abuse (excluding tobacco use or use of medical or recreational marijuana) within the 12 months prior to Screening or evidence of such abuse, in the opinion of the Investigator.
8. Limited life expectancy (less than 6 months) in the opinion of the Investigator.
9. Females who are known to be pregnant or are breast-feeding during Screening or are planning to become pregnant and breastfeeding during the study period.
10. Evidence of a clinically active infection requiring antibiotics at Randomization.
11. Unable to comply with study requirements or in the opinion of the Investigator, not clinically stable to participate in the study.
12. Use of an investigational medication or participation in an investigational study within 30 days prior to Day 1.
13. Patients with a scheduled date for receipt of living donor kidney transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Block, MD, Principal Investigator — USRC Kidney Research
Locations (20):
- United States (20):
  - Arkansas Nephrology & Hypertension Clinic, Pine Bluff, Arkansas
  - Balboa Research SMO, Chula Vista, California
  - Balboa Research SMO, El Centro, California
  - Balboa Research SMO, Escondido, California
  - Balboa Research SMO, La Mesa, California
  - Balboa Research SMO - Kearney Mesa, San Diego, California
  - Rocky Mountain Kidney Care, Lone Tree, Colorado
  - Associates in Nephrology, Fort Myers, Florida
  - Dialysis Clinic, Inc., Albany, Georgia
  - Nephrology and Hypertension Specialists, PC, Dalton, Georgia
  - Major Health Partners, Shelbyville, Indiana
  - Kidney Associates of Kansas City, Kansas City, Missouri
  - Nephrology-Hypertension Associates of Central NJ, South River, New Jersey
  - High Desert Nephrology Associates, Gallup, New Mexico
  - Nephrology Associates of Western NY, Amherst, New York
  - Spartanburg Nephrology Associates, Spartanburg, South Carolina
  - Dialysis Clinic, Inc., Knoxville, Tennessee
  - South Texas Renal Care Group, Live Oak, Texas
  - South Texas Renal Care Group, San Antonio, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, double-blind, placebo-controlled clinical trial to assess the effect of ferric citrate on the time to a composite endpoint of initiation of maintenance dialysis or all-cause mortality compared with placebo in adults with advanced chronic kidney disease.
Pre-assignment Details: A total of 289 patients were randomized 1:1 to receive ferric citrate (n=144) or placebo (n=145).
Period: Overall Study
Arm/Group | Ferric Citrate | Placebo
Started | 144 | 145
Received Day 1 Dose | 138 | 136
Completed | 88 | 77
Not Completed | 56 | 68

BASELINE CHARACTERISTICS:
Population: This patient population includes those patients that were consented, eligible to be enrolled, randomized, and received a Day 1 dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferric Citrate | Placebo | Total
Number analyzed (Participants) | 138 | 136 | 274
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Total number of patients should be 274: (Ferric citrate (N=138) and Placebo (N=136).
  years | 66.3 (13.1) | 68.2 (12.9) | 67 (13)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Total number of patients should be 274: (Ferric citrate (N=138) and Placebo (N=136).
  Participants
    Female | 79 | 71 | 150
    Male | 59 | 65 | 124
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Total number of patients should be 274: (Ferric citrate (N=138) and Placebo (N=136).
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 24 | 21 | 45
    White | 94 | 97 | 191
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 20 | 18 | 38
Comorbid conditions at baseline [Count of Participants; unit: Participants] — Population: Total number of patients should be 274: (Ferric citrate (N=138) and Placebo (N=136).
  Participants
    Atherosclerotic cardiovascular disease | 41 | 55 | 96
    Congestive heart failure | 20 | 30 | 50
    Diabetes | 92 | 86 | 178

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving a Composite Endpoint of Initiation of Maintenance Dialysis or All-cause Mortality
Description: Number of participants achieving a composite endpoint of initiation of maintenance dialysis or all-cause mortality
Time Frame: 9 months
Population: Full analysis set which consists of randomized patients who received one or more doses of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ferric Citrate | Placebo
Number analyzed (Participants) | 138 | 136
Participants | 35 | 46
Statistical Analysis 1: Comparison: Ferric Citrate vs Placebo; Test type: Non-Inferiority — The study planned to enroll 400 patients (200 patients in each treatment arm) to achieve 90% power to detect a hazard ratio (HR) of 0.60 for the primary composite endpoint, with differences between treatment groups assessed using a 2-sided alpha of <0.05; p = .1602, Regression, Cox; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.46 to 1.14]

2. Secondary Outcome: Hospitalization Events Reported as a Serious Adverse Event (SAE) (Excluding Disease-related Hospitalization [e.g., Dialysis Access Placement, Dialysis Initiation, Kidney Transplant] and Elective Procedures)
Description: Number of hospitalization events reported as a serious adverse event (SAE) (excluding disease-related hospitalization [e.g., dialysis access placement, dialysis initiation, kidney transplant] and elective procedures)
Time Frame: 9 months
Population: Full analysis set population which consists of all randomized patients who received one or more doses of study drug.
Measure: Mean (Standard Deviation); unit: Number of hospitalizations per patient
Arm/Group | Ferric Citrate | Placebo
Number analyzed (Participants) | 138 | 136
Number of hospitalizations per patient | 1.1 (2.4) | 2.5 (9.4)

3. Secondary Outcome: Component of Primary - Initiation of Maintenance Dialysis
Description: Component of Primary - Number of participants initiating maintenance dialysis
Time Frame: 9 months
Population: Full analysis set population which consists of all randomized patients who received one or more doses of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ferric Citrate | Placebo
Number analyzed (Participants) | 138 | 136
Participants | 24 | 29
Statistical Analysis 1: Comparison: Ferric Citrate vs Placebo; Test type: Other; p = .30, Regression, Cox; Hazard Ratio (HR) = 0.78, Standard Error of Mean .2392

4. Secondary Outcome: Component of Primary - All-Cause Mortality
Description: Component of Primary - Number of patients reaching endpoint of all-cause mortality.
Time Frame: 9 months
Population: Full analysis set population which consists of all randomized patients who received one or more doses of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ferric Citrate | Placebo
Number analyzed (Participants) | 138 | 136
Participants | 1 | 4
Statistical Analysis 1: Comparison: Ferric Citrate vs Placebo; Test type: Other; p = 0.17, Regression, Cox; Hazard Ratio (HR) = 0.35, Standard Error of Mean 0.8295

ADVERSE EVENTS:
Time Frame: Serious Adverse Events and Adverse Events of Special Interest were collected from initiation of study drug treatment through the 10 months.
Description: Only Serious Adverse Events and Adverse Events of Special Interest (Iron Overload and Clinically Significant Hypophosphatemia) were collected.
Arm/Group | Ferric Citrate | Placebo
All-Cause Mortality (participants affected / at risk) | 2/138 | 6/136
Serious Adverse Events (participants affected / at risk) | 33/138 | 43/136
Other Adverse Events (participants affected / at risk) | 0/138 | 0/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ferric Citrate (N=138) | Placebo (N=136)
Anaemia (Blood and lymphatic system disorders) | 1 | 4
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 6 | 6
Cardiac arrest (Cardiac disorders) | 1 | 4
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Retinal artery occlusion (Eye disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Cardiac death (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Sepsis (Infections and infestations) | 3 | 1
Pyelonephritis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 3
Skin infection (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1
Emphysematous cystitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 2
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 3
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 5
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
End stage renal disease (Renal and urinary disorders) | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypertension (Vascular disorders) | 1 | 0
Malignant hypertension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication or disclosure of study results will be permitted, except under the terms and conditions of a separate, written agreement between Investigator-Sponsor and the Investigator and/or the Investigator's institution. The Investigator-Sponsor will have the opportunity to review and approve all proposed abstracts, manuscripts, or presentations regarding this study prior to submission for publication/presentation.

DOCUMENTS (2):
  • Study Protocol (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT05085275/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/75/NCT05085275/SAP_001.pdf